CLINICAL TRIAL: NCT04852068
Title: A Randomized, Blinded, and Similar Vaccine-controlled Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of the 5-dose Program and 4-dose (2-1-1) Program of Freeze-dried Human Rabies Vaccine (Vero Cells)
Brief Title: A Clinical Trial of Freeze-dried Human Rabies Vaccine (Vero Cells)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2020-Rab01
Record Dates: First submitted 2021-04-12; First posted 2021-04-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Rabies Vaccine Adverse Reaction; Safety and Efficacy

STUDY DESIGN:
Intervention Model Description: Similar vaccine control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Investigational Vaccine - 5-dose program (Experimental): Freeze-dried human rabies vaccine (Vero cells), 0.5ml after reconstitution, with a titer of not less than 2.5IU, Anhui Zhifeilongkoma Biopharmaceutical Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (Vero cells) Zhifeilongkoma - 5-dose program
- Investigational Vaccine - 4-dose program (Experimental): Freeze-dried human rabies vaccine (Vero cells), 0.5ml after reconstitution, with a titer of not less than 2.5IU, Anhui Zhifeilongkoma Biopharmaceutical Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (Vero cells) Zhifeilongkoma - 4-dose program
- Control vaccine - 5-dose program (Active Comparator): Freeze-dried human rabies vaccine (Vero cells), 0.5ml after reconstitution, titer not less than 2.5IU, Liaoning Chengda Biological Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (Vero cells) Chengda - 5-dose program
- Control vaccine - 4-dose program (Active Comparator): Freeze-dried human rabies vaccine (Vero cells), 0.5ml after reconstitution, titer not less than 2.5IU, Liaoning Chengda Biological Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (Vero cells) Chengda - 4-dose program

INTERVENTIONS:
Biological: Freeze-dried human rabies vaccine (Vero cells) Zhifeilongkoma - 5-dose program — Inoculate 1 dose of Investigational vaccine each on 0, 3, 7, 14, 28 days, by intramuscular injection of deltoid muscle of upper arm
  Arms: Investigational Vaccine - 5-dose program
Biological: Freeze-dried human rabies vaccine (Vero cells) Zhifeilongkoma - 4-dose program — Inoculate 1 dose of Investigational vaccine each on both arms on day 0, and 1 dose each on day 7 and 21, by intramuscular injection of deltoid muscle of upper arm
  Arms: Investigational Vaccine - 4-dose program
Biological: Freeze-dried human rabies vaccine (Vero cells) Chengda - 5-dose program — Inoculate 1 dose of control vaccine each on 0, 3, 7, 14, 28 days, by intramuscular injection of deltoid muscle of upper arm
  Arms: Control vaccine - 5-dose program
Biological: Freeze-dried human rabies vaccine (Vero cells) Chengda - 4-dose program — Inoculate 1 dose of control vaccine each on both arms on day 0, and 1 dose each on day 7 and 21, by intramuscular injection of deltoid muscle of upper arm
  Arms: Control vaccine - 4-dose program

SUMMARY:
This clinical trial is carried out in two phases. The first phase adopts an open design, and the second phase adopts a randomized, blinded, and similar vaccine-controlled non-inferiority trial design.

The first stage: According to the order of two age groups of 18-60 years old and 10-17 years old, 40 cases were enrolled in each age group (20 persons for the 5-dose program and 20 for the 4-dose program). Subjects in the 5-dose group received 1 dose of test vaccine on 0, 3, 7, 14, and 28 days each. Subjects in the 4-dose group received 1 dose each on both arms on day 0, and 1 dose on day 7 and day 21 each. All subjects in the first stage were only observed for safety and were followed up to 6 months after the entire course of vaccination.

The second stage: the total number of enrolled 2400 cases, 10-60 years old, the 4-dose program group and the 5-dose program group of the test vaccine, the 4-dose program group and the 5-dose program group of the control vaccine according to the random ratio 1:1:1:1. Among the total number of participants, 1680 cases (420 cases per group) were simultaneously observed for immunogenicity and safety, and the remaining 720 subjects (180 cases per group) only underwent safety observation. 800 subjects (200 cases in each group) received 6-month immune persistence observation after full vaccination, and 400 subjects in the test vaccine group received 12 months immune persistence observation after full vaccination.

In the second stage, 1680 subjects were collected before the immunization, 7 days after the first dose, 14 days after the first dose, and 14 days after the full vaccination to test rabies virus antibodies to evaluate the immunogenicity of the test vaccine. 800 subjects were in the whole process Immune persistent blood sampling was performed 6 months after vaccination, and subjects in the test vaccine group were further subjected to immune persistent blood sampling 12 months after the full course of vaccination to evaluate immune durability. Collect all AEs within 30 minutes after each dose, AEs from 0-7 days, all non-collective AEs from the first dose to 30 days after the full course of vaccination, and all serious AEs from the first dose to 6 months after the full course of vaccination Adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-60 on the day of enrollment, able to provide legal identification
* Subjects and/or their guardians voluntarily agree to participate in the study and sign an adult informed consent form or a minor's informed consent form
* Subjects and/or their legal guardians have the ability to understand (non-illiterate) research procedures and participate in all planned follow-ups
* On the day of enrollment, the axillary body temperature of people aged 14 and under was <37.5℃, and the axillary body temperature of people over 14 years of age was <37.3℃
* Female subjects of childbearing age were not breast-feeding at the time of enrollment, were not pregnant (the urine pregnancy test was negative before vaccination (on the day)), had no pregnancy plan within 2 months after enrollment, and agreed to take effective measures within 2 months after enrolling in the study Contraceptive measures

Exclusion Criteria:

* Have a history of rabies vaccination or use of rabies virus passive immunization preparations
* A history of bites by mammals (such as dogs, cats, etc.) within 1 year before the first dose of vaccination (wound skin damage)
* Previous vaccination has a history of severe allergies to any vaccine component that requires medical intervention: such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis, severe urticaria, etc.
* Within 3 days before vaccination, acute febrile disease (body temperature under armpit>38.5℃) or in the acute onset of chronic disease, or taking antipyretic, analgesic, and anti-allergic drugs
* Have received blood/blood-related products or immunoglobulins within 3 months before the first dose of vaccination; or plan to use such products within 1 month after the last dose of vaccination
* Get any vaccine within 14 days before the first dose of vaccination
* Any condition (such as splenectomy) caused asplenia or functional asplenia
* Has been diagnosed with congenital or acquired immunodeficiency (HIV), or received immunosuppressive therapy within 3 months
* Severe congenital malformations or autoimmune (hereditary) diseases, serious chronic diseases (including but not limited to: heart disease, kidney disease, diabetes with comorbidities, allergic constitution, Guillain-Barre syndrome, etc.), evaluated by the investigator that it may affect research evaluation
* People with a history or family history of convulsions, epilepsy, encephalopathy, and psychosis (including but not limited to: congenital brain hypoplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral obstruction, brain nerve tissue damage caused by infection, chemical drug poisoning, etc.)
* There are contraindications for intramuscular injection (diagnosed as any coagulation disorder or receiving anticoagulant treatment)
* Are participating in other research or unregistered products (drugs, vaccines or devices, etc.) clinical research, or plan to participate in other clinical research before the end of this clinical research
* The researcher believes that the subject has any conditions that may interfere with the evaluation of the research purpose

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2480 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Antibody positive conversion rate - Immunogenicity endpoint | 14 days after the first dose of vaccination
  Antibody positive conversion rate of the test group and the control group of the pre-immune antibody-negative population
Geometric mean concentration - Immunogenicity endpoint | 14 days after the first dose of vaccination
  Geometric mean concentration of the test group and the control group of the pre-immune antibody-negative population
Incidence of Adverse Events [Safety and Tolerability] | within 30 minutes after each dose of vaccination; the first dose of vaccination to 30 days after the full course of vaccination
  Incidence of Adverse Events
Incidence of Serious Adverse Events [Safety and Tolerability] | The first dose of vaccination to 6 months after the full course of vaccination
  Incidence of Serious Adverse Events

SECONDARY OUTCOMES:
Antibody positive conversion rate - Immunogenicity endpoint | 7 days after the first dose of vaccination; 14 days, 6 months, 12 months after the full vaccination
  Antibody positive conversion rate
Geometric mean concentration - Immunogenicity endpoint | 7 days after the first dose of vaccination; 14 days, 6 months, 12 months after the full vaccination
  Geometric mean concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No